CLINICAL TRIAL: NCT05265650
Title: Phase Ib/II Open-label Clinical Study of Intratumoral Administration of BO-112 in Combination With Radiotherapy and Nivolumab in Patients With Metastatic PD- 1/PD-L1 Refractory Non-small Cell Lung Cancer
Brief Title: Study of BO-112 With Radiotherapy and Nivolumab for Metastatic Refractory NSCLC
Acronym: Noelia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Highlight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BORT-112
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Non-Small Cell Lung Cancer Metastatic
Keywords: BO112; Intratumoral; Immunotherapy; NSCLC
MeSH Terms: interventions — BO-112; Radiosurgery; Nivolumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is a phase Ib/II study with one single treatment arm (BO-112 in combination with SABR and nivolumab)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Treatment Arm (Experimental): Treatment will consist of IT administrations of BO-112 in combination with ablative radiotherapy (SABR) and concurrent with systemic administration of nivolumab in patients with metastatic PD-1/PD-L1-refractory NSCLC.
  In the initial cohort A, BO-112 will be IT injected on a weekly basis during the first cycle on the accessible lesions, and every 2 weeks thereafter. The minimum dose to be injected per visit is 1 mg (unless injected lesion in case of response, if solitary, becomes smaller than 1.5 cm) and the maximum dose is 2 mg (3.4 mL), distributed in the different lesions.
  Stereotactic ablative radiotherapy (SABR) will be initiated on week 3.
  In the cohort B, BO-112 and SABR will be administered as described previously.
  Nivolumab will be administered at the dose of 240 mg every 2 weeks in both cohorts, starting at cycle 4 (week 7) in cohort A and at cycle 3 (week 5) in cohort B.
  Interventions: Drug: BO-112 in combination with ablative radiotherapy (SABR) and nivolumab; Procedure: Tissue Biopsies

INTERVENTIONS:
Drug: BO-112 in combination with ablative radiotherapy (SABR) and nivolumab — Study treatment will consist of BO-112 IT injections in combination with IV nivolumab infusions and SABR to accessible metastases.
  Other Names: BO-112 with radiotherapy and nivolumab
Procedure: Tissue Biopsies — Four research biopsies will be taken from accessible injected lesions, at the time of the IT injection of BO-112.

SUMMARY:
This is a study of repeated IT administrations of BO-112 in combination with ablative radiotherapy (SABR) and concurrent nivolumab in patients with metastatic PD-1/PD-L1-refractory NSCLC.

DETAILED DESCRIPTION:
This is a phase Ib/II study to evaluate feasibility-efficacy of repeated IT administrations of BO-112 in combination with ablative radiotherapy (SABR) and concurrent with systemic administration of nivolumab in patients with metastatic PD-1/PD-L1-refractory NSCLC.

To be eligible, all patients must have metastatic NSCLC with at least one accessible lesion amenable to IT BO-112 injection and radiotherapy administration. The study will include an initial cohort A using a standard "3+3" design to determine the safety profile of SABR in combination with BO-112 and nivolumab, which will start on cycle 4 (week 7) and a cohort B, with the same combination but with nivolumab starting on cycle 3 (week 5).

In the initial cohort A, BO-112 will be IT injected on a weekly basis during the first cycle on the accessible lesions, and every 2 weeks thereafter. On the liver, the maximum frequency for IT injection will be every 2 weeks since the first administration. After the first cycle, BO-112 will continue to be IT injected every 2 weeks on the previously treated lesions provide they are still injectable. A maximum of 2 hepatic lesions will be treated with BO-112 at each cycle and a maximum of 5 multisite tumoral lesion in total. The minimum dose to be injected per visit is 1 mg (unless injected lesion in case of response, if solitary, becomes smaller than 1.5 cm) and the maximum dose is 2 mg (3.4 mL), distributed in the different lesions. Distribution of volume of injection will be determined based on the size of lesion to be injected. Stereotactic ablative radiotherapy (SABR) will be initiated on week 3. Patients will be evaluated for DLTs until 28 days after the first dose of nivolumab.

In cohort B, BO-112 and SABR will be administered as described previously.

Nivolumab will be administered at the dose of 240 mg every 2 weeks in both cohorts, starting at cycle 4 (week 7) in cohort A and at cycle 3 (week 5) in cohort B.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. ≥18 years of age
3. Diagnosis of histologically confirmed metastatic NSCLC (histologic confirmation of a NSCLC tumor is acceptable if accompanied by radiographic evidence of metastatic disease).
4. At least 1 accessible metastasis of minimum 20 mm in diameter that is suitable for percutaneous IT injection of BO-112. For liver metastasis IT injection, the lesion to be treated cannot infiltrate the main hepatic vessels (including, but not limited to, absence of tumor infiltration into the main portal vein, hepatic vein, or vena cava) and must be amenable to be biopsied. The irradiated and injected site must be accessible to tumor biopsy.
5. Presence of at least 1 measurable lesion according to RECIST v. 1.1. Note: this may be the metastasis selected for injection if it is the only measurable lesion present.
6. Prior resection of metastatic disease is allowed if completed more than 6 months previous to study enrollment and at the time of study entry there is progressive disease.
7. Patients must be refractory to anti-PD-1, or anti-PD-L1 inhibitors. Subjects who have received prior anti-PD-1/PD-L1 therapies must have received at least 4 months of treatment. Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided at least 2.5 half-lives (30 days) have elapsed from the last dose of anti-CTLA-4 to the first dose of nivolumab and there was no history of severe immune-mediated adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3 and 4). Subjects with EGFR or ALK genomic tumor aberrations with progression on approved therapy for these aberrations are eligible.
8. Participant must be candidate for SABR to at least 1 lesion with no more than 5 irradiated metastases in total. Maximum of 3 metastases to be irradiated in any one organ are allowed.
9. Evaluation by a radiation oncologist within 21 days prior to study registration, including imaging workup to document metastases.
10. Irradiation by SABR should not include metastases located within 3 cm of the previously irradiated structures:

    * Spinal cord previously irradiated to >40 Gy.
    * Brachial plexus previously irradiated to >50 Gy.
    * Small intestine, large intestine, or stomach previously irradiated to >45 Gy.
    * Brainstem previously irradiated to >50 Gy.
    * Lung previously irradiated with prior V20 Gy >30%.
11. Have performance status of 0 or 1 on the ECOG Performance Scale.
12. Adequate hematologic and end-organ function defined by the following laboratory results obtained at screening and at Visit 1 prior to the first dose of study treatment:

    * ANC ≥1.5 × 109/L.
    * Platelet count ≥100 × 109/L.
    * Hemoglobin ≥9.0 g/dL.
    * AST and ALT ≤2.5 × ULN (5 × ULN if presence of liver metastases).
    * Serum total bilirubin <2 × ULN (if known Gilbert's syndrome, serum bilirubin level <3 × ULN).
    * Prothrombin time (PT) (or international normalized ratio [INR]) within normal limits and activated partial prothrombin time (aPTT) within normal limits.
    * Serum creatinine <1.5 × ULN or creatinine clearance ≥30 mL/min (calculated per cockcroft formula).
13. Female participants of childbearing potential should have a negative urine or serum pregnancy test within 10 days of initiating study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Female participants of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. (Appendix 7). Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.
15. Male participant should agree to use an adequate method of contraception starting and refrain from sperm donation with the first dose of study therapy through 6 months after the last dose of study therapy.
16. HIV infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

    * Participants on ART must have a CD4+ T-cell count >350 cells/mm3 at time of screening.
    * Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening.
    * Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (Day 1).
17. Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.

    Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
18. Hepatitis B screening tests are not required unless:

    * Known history of HBV infection.
    * As mandated by local health authority.
19. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

    Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.
20. Hepatitis C screening tests are not required unless:

    * Known history of HCV infection.
    * As mandated by local health authority.
21. Able and willing to comply with study and follow-up procedures.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

1. Prior treatment with any Toll-like receptor (TLR) agonist or sting agonist.
2. Chemotherapy, definitive (curative) radiation, or biological cancer therapy within 4 weeks prior to the first dose of study treatment. Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. If the participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
3. Palliative radiotherapy (≤2 weeks of radiotherapy) within 1 week of start of study treatment. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
4. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases. Patients with a history of treated CNS metastases are eligible, providing all of the following criteria are met:

   * Measurable disease, per RECIST v. 1.1, must be present outside the CNS.
   * The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
   * Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
   * There is no evidence of interim radiological progression for at least 4 weeks between completion of CNS-directed therapy and the screening brain scan.
   * The patient has clinical stability from the neurological point of view and doesn´t require corticosteroids as therapy for CNS disease for at least 14 days. Anti-convulsant therapy at a stable dose is permitted.
5. History of leptomeningeal disease.
6. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
7. Life expectancy of <12 weeks.
8. Active infection requiring systemic therapy within 1 week of start of study treatment.
9. Serious medical comorbidities precluding radiotherapy. These include, but are not limited to, the following:

   * Interstitial lung disease in patients requiring thoracic radiation.
   * Crohn's disease in patients where the GI tract will receive radiotherapy, or ulcerative colitis where the bowel will receive radiotherapy.
   * Connective tissue disorders such as lupus or scleroderma.
   * Known genetic disorders associated with increased toxicity to radiation therapy (e.g., ataxia telangiectasia).
10. For patients with liver metastases:

    * Moderate/severe liver dysfunction (Child Pugh B or C).
    * Liver metastasis(es) with macroscopic tumor infiltration into the main portal vein, hepatic vein, or vena cava.
11. Substantial overlap with a previously treated radiation volume:

    * Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein.
    * For patients treated with radiation previously, biological effective dose calculations should be used to equate previous doses to the tolerance doses listed in the technical radiotherapy manual. All such cases must be discussed with the Medical Monitor and the responsible radiotherapy investigator at the site.
    * Lesions that have been treated with radiotherapy within the last 6 months should not be radiated.
12. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Use of an indwelling catheter (e.g., PleurX®) is allowed.
13. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

    Note: History of radiation pneumonitis <grade 3 in the radiation field (fibrosis) is permitted.
14. Active autoimmune disease that required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
15. Receiving systemic immunosuppressive therapy within 28 days before enrolment with the exceptions of intranasal, topical, and inhaled corticosteroids or oral corticosteroids at physiological doses not exceeding 10 mg/day of prednisone or equivalent.
16. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
17. For WOCBP: pregnancy or a positive urine pregnancy test (e.g., within 72 hours) prior to treatment; or breastfeeding. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
18. Any other medical condition which would impact the safety of the subject or interfere with the subject's ability to comply with the study and follow-up procedures, in the opinion of the investigator.
19. Has received a live vaccine within 28 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed. COVID vaccines may be administered, but always allowing a wash out period of at least 72 hours between vaccine and BO-112 dose.
20. Is currently participating or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment (subjects who are in a follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent).
21. Has had an allogenic tissue/solid organ transplant.
22. Significant bleeding event within the last 12 months that places the patient at risk for intrahepatic IT injection procedure based on Investigator assessment.
23. Contraindications to tumor biopsy and IT injections of BO-112, such as coagulopathy, therapeutic dose anticoagulant treatment and treatment with long-acting agents. Anticoagulant or anti-platelet medication that cannot be interrupted prior to BO-112 IT injection, including:

    * Aspirin that cannot be discontinued for 7 days prior to BO-112 IT injection.
    * Coumadin that cannot be discontinued for 7 days prior to BO-112 IT injection.
    * Low molecular weight heparin (LMWH) that cannot be discontinued >24 hours prior to BO-112 IT injection.
    * Unfractionated heparin (UFH) that cannot be discontinued >4 hours prior to BO-112 IT injection.
    * Oral direct thrombin inhibitor (dabigatran) or direct Factor Xa inhibitor (rivaroxaban, apixaban, and edoxaban) that cannot be discontinued for 4 days prior to BO-112 IT injection.

Note: LMWH or UFH may be used to transition patients on and off of the above anti-coagulants (if deemed appropriate by the treating physician) prior to BO-112 IT injection as long as the last dose of LMWH is administered >24 hours prior to treatments and last dose of UFH is administered >4 hours prior to treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events and Serious Adverse Events | Throughout study completion, an average of 1 year
  Number and proportion of subjects with TEAEs with severity ≥ Grade 3 (NCI-CTCAE v. 5.0)

SECONDARY OUTCOMES:
Number and Proportion of Subjects with TEAEs Grade ≥3 | Throughout study completion, an average of 1 year
  Number and proportion of subjects with study treatment-related TEAEs Grade ≥3, number and proportion of subjects with TEAEs (any grade); number and proportion of subjects with related TEAEs (any grade).
Efficacy: Progression-free survival (PFS) | Throughout study completion, an average of 1 year
  t Time from C1D1 to the first occurrence of disease progression or death from any cause
Efficacy: ORR, DCR | Throughout study completion, an average of 1 year
  ORR based on the best overall response (BOR); disease control rate (DCR = CR, PR and SD of at least 12 weeks duration) on the global tumor assessment in ITT population.
  * DCR = iCR, iPR + iSD of at least 12 weeks duration) in ITT population.
  * Overall survival rate at 12 months.
Tolerability: study discontinuations | Throughout study completion, an average of 1 year
  Number of study discontinuations due to related TEAE.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Rodriguez, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No